CLINICAL TRIAL: NCT03711760
Title: Telepsychology Intervention for Individuals With Spinal Cord Injury and Depression
Brief Title: Telepsychology in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Collaborators: University of California, San Francisco (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC170243; SC170243 (Other Grant/Funding Number: CDMRP-eBRAP Log Number)
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Depression
Keywords: telepsychology; spinal cord injuries; depression; cognitive behavioral therapy
MeSH Terms: conditions — Spinal Cord Injuries; Depression | interventions — Mental Health Teletherapy

STUDY DESIGN:
Intervention Model Description: single center, blinded assessor, controlled, randomized, intention to treat.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): telepsychology treatment
  Interventions: Behavioral: telepsychology
- usual care (No Intervention): standard of care

INTERVENTIONS:
Behavioral: telepsychology — CBT delivered by telepsychology
  Arms: intervention

SUMMARY:
This study will determine the effectiveness of tele-psychology in treating persons with spinal cord injury (SCI) with depressed mood in the early period post-rehabilitation discharge. Depression among individuals with SCI is the most common psychological condition following an injury; 22% of civilians with SCI and 28% of veterans with SCI experience depression after injury, which is higher than the able-bodied population (Williams 2015; Ullrich 2014). Individuals with SCI face many barriers in receiving psychotherapy, such as lack of accessible transportation, unfamiliarity with community resources, or stigma associated with seeking treatment for depression, which this project aims to address. Cognitive behavior therapy (CBT), which helps people develop different ways of thinking and behaving to reduce their psychological distress, will be provided via iPad FaceTime by a psychologist with expertise in working with persons with SCI.

The objectives of the proposed project are to reduce depressive symptoms, decrease associated symptoms of anxiety, and to improve satisfaction with life with CBT provided via tele-psychology. The secondary objective is to show intermediate efficacy of tele-psychology in persons with SCI with depressed mood.

DETAILED DESCRIPTION:
I. Rationale / Objectives This study will determine the effectiveness of tele-psychology in treating persons with spinal cord injury (SCI) with depressed mood in the early period post-rehabilitation discharge. Depression among individuals with SCI is the most common psychological condition following an injury; 22% of civilians with SCI and 28% of veterans with SCI experience depression after injury, which is higher than the able-bodied population (Williams 2015; Ullrich 2014). Individuals with SCI face many barriers in receiving psychotherapy, such as lack of accessible transportation, unfamiliarity with community resources, or stigma associated with seeking treatment for depression, which this project aims to address. Cognitive behavior therapy (CBT), which helps people develop different ways of thinking and behaving to reduce their psychological distress, will be provided via iPad FaceTime by a psychologist with expertise in working with persons with SCI.

The objectives of the proposed project are to reduce depressive symptoms, decrease associated symptoms of anxiety, and to improve satisfaction with life with CBT provided via tele-psychology. The secondary objective is to show intermediate efficacy of tele-psychology in persons with SCI with depressed mood.

II. Impact CBT via iPad FaceTime is expected to be a convenient and effective treatment for depression after SCI with short-term (14-week post-discharge) and intermediate (26-week post-discharge) benefits. This project would impact individuals with SCI, post-discharge from rehabilitation, through the provision of an innovative treatment for depression, easing the transition back to their home and community. Furthermore, CBT treatment will be provided in the comfort and privacy of the participant's home, therefore combating stigma, as well as physical and transportation-associated barriers. CBT via FaceTime does pose a potential confidentiality risk, but the study team will stress that both parties choose a location (i.e. private office for the psychologist and a private room at home for the participant) that will minimize this risk. Prior studies have shown a beneficial effect of CBT provided with tele-psychology among other populations. Telemedicine is rapidly advancing within the field of medicine; however, its impact on persons with SCI and the use of tele-psychology are not yet widespread. This proposed study aims to close this gap and can determine whether CBT via iPad improves mood and quality of life (as measured by satisfaction with life) and can assess if tele-psychology is an effective and replicable method for providing psychological care. With evidence from this study elucidating the effectiveness of tele-psychology utilizing rapidly advancing technology, tele-psychology for individuals with SCI may become as usual and routine as in-person psychological treatment within several years.

III. Contribution This project provides an innovative approach to treating depression and an exciting opportunity to understand the treatment effects of our proposed tele-psychological intervention for individuals with SCI. CBT treatment provided via iPad FaceTime tele-psychology for depression is a novel approach that can easily be disseminated to other SCI centers and community hospitals. Hence, medical teams will have an alternative option to consider during the discharge planning stages of rehabilitation and during their transition to home.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening Inclusion Criteria:

* Adults 18 years or older with traumatic or non-traumatic SCI at any level of injury
* Individuals with acute SCI being discharged to or residing in a private residence in the state of California
* Within one year of date of injury

Tele-psychology (full study) Inclusion Criteria:

* Mild to moderate depression (PHQ-9 total score between 5-14)
* Intact cognitive status (i.e., full scale MoCA ≥ 25). Potential subjects being screened remotely or who cannot complete the motoric components of the MoCA will be screened with the MoCA Blind (required score ≥ 17)

Exclusion Criteria:

Pre-screening Exclusion Criteria:

* Medically unstable as determined by the subject's treating physician or a review of medical records (e.g. pneumonia)
* Acute psychosis
* Incapable of giving informed consent
* Inability to comprehend written or oral English
* For Non-County of Santa Clara Residents: Inability to identify a treating physician to the study team. (* Please contact the study team if you are not sure who your treating physician may be)

Tele-psychology (full study) Exclusion Criteria:

* Endorsement of suicidality on the PHQ-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Baseline, 12 weeks, 24 weeks
  The Patient Health Questionnaire - 9 is a 9-item tool for assessment of depression severity. It has a total scoring range of 0 to 27, and a higher score signifies more severe depression.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder-7 | Baseline, 12 weeks, 24 weeks
  The Generalized Anxiety Disorder Instrument is a 7-item tool for assessment of anxiety severity. It has a total scoring range of 0 to 21, and a higher score signifies more severe anxiety.
Change in Satisfaction with Life Scale | Baseline, 12 weeks, 24 weeks
  The Satisfaction with Life Scale is a 5-item tool for assessing life satisfaction and subjective quality of life. It has a total scoring range of 7-35, and a higher score signifies better satisfaction with life.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Shem, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rehabilitation Research Center — https://www.scvmc.org/health-care-services/rehabilitation/rehabilitation-research-center/research-projects